CLINICAL TRIAL: NCT05869058
Title: Development and Improvement of a Deep Convolutional Neural Network for Detection and Assessing the Perfusion of Parathyroid Gland During Endoscopic Thyroidectomy
Brief Title: DCNN Developed for Detection and Assessing the Perfusion of PTG
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-177-01
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: a deep convolutional neural network — a deep convolutional neural network developed for detection and assessing the perfusion of parathyroid gland during endoscopic thyroidectomy

SUMMARY:
Since the anatomical location and appearance of the parathyroid gland (PTG) vary, detection of the PTG and preserving the blood supply are among the difficulties encountered during a thyroidectomy procedure. We are planning to train a deep convolutional neural network based on a larger sample of endoscopic images to develop a model to assist surgeons in detection of PTG during endoscopic thyroidectomy. Furthermore, we would like to train a DCNN to predict blood perfusion based on endoscopic images comparing to indocyanine green fluorescence angiography as reference standard, and assess the performance of DCNN in predicting postoperative hypoparathyroidism.

DETAILED DESCRIPTION:
Since the anatomical location and appearance of the parathyroid gland (PTG) vary, detection of the PTG and preserving the blood supply are among the difficulties encountered during a thyroidectomy procedure. Resection of the PTG by mistake or interruption of the blood supply may lead to transient or permanent hypoparathyroidism, which would require short-term or lifelong calcium and/or vitamin D supplement. We are planning to train a deep convolutional neural network based on a larger sample of endoscopic images to develop a model to assist surgeons in detection of PTG during endoscopic thyroidectomy. Although several researchers indicated that indocyanine green fluorescence angiography could be used to assess the perfusion of the PTG intraoperatively, it may cause allergic reaction and need repetitive injection. Therefore, we would like to train a DCNN to predict blood perfusion based on endoscopic images comparing to indocyanine green fluorescence angiography as reference standard, and assess the performance of DCNN in predicting postoperative hypoparathyroidism. This research may lead to the development of endoscopic modules in PTG detection and PTG perfusion prediction to reduce postoperative hypoparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* The patients who undergo endoscopic thyroidectomy

Exclusion Criteria:

* hyperparathyroidism
* hypoparathyroidism
* neck surgery history
* cervical radiotherapy history

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients, who choose to undergo endoscopic thyroidectomy due to thyroid diseases and have no history of hyperparathyroidism, hypoparathyroidism, neck surgery and cervical radiotherapy, are candidates of our study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve | 3 years
  Area Under the Receiver Operating Characteristic Curve

CONTACTS AND LOCATIONS:
Overall Officials: Peiliang Lin, M.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China